CLINICAL TRIAL: NCT05048550
Title: Can Provision of Near Vision Glasses as an Early Intervention Improve Visual and Developmental Outcomes in Children With Perinatal Brain Insult? A Feasibility Study.
Brief Title: Babies in Glasses; a Feasibility Study.
Acronym: BiG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University College London Hospitals (Other); University College, London (Other); University of Reading (Other); University of Bristol (Other); University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18BA36
Record Dates: First submitted 2021-06-24; First posted 2021-09-17 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Cerebral Visual Impairment; Refractive and Accommodative Disorders; Hypoxic-Ischemic Encephalopathy; Premature Birth
Keywords: Cerebral Visual Impairment; CVI; Visual Processing Disorder; Visual Perceptual Deficits; VPD; Accommodative Disorders; Hypo-accommodation; Accommodative lag; Hypoxic Ischaemic Encephalopathy; Premature Birth; Near Vision Glasses; Spectacle correction; Refractive correction; Refractive Error; Early spectacle correction; Spectacles; Glasses; Perinatal Brain Insult; Brain Injury; Neurodevelopment; Infant; Baby; Functional broadband Near Infrared Spectroscopy; fBNIRS
MeSH Terms: conditions — Blindness, Cortical; Hypoxia-Ischemia, Brain; Premature Birth; Refractive Errors; Brain Injuries

STUDY DESIGN:
Intervention Model Description: This is a single-centre randomised interventional study; a 3-arm parallel group, open-label clinical feasibility trial for a definitive RCT with equal arm allocation and a superiority design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A (control) (No Intervention): First visit assessments at 8 weeks corrected gestational age. No glasses prescribed.
- B1 (intervention) (Experimental): First visit assessments at 8 weeks corrected gestational age. Full time spectacle wear prescribed.
  Interventions: Device: Near vision spectacles
- B2 (intervention) (Experimental): First visit assessments at 16 weeks corrected gestational age. Full time spectacle wear prescribed.
  Interventions: Device: Near vision spectacles

INTERVENTIONS:
Device: Near vision spectacles — Near vision spectacles prescribed for full time wear (Add+3.00DS to the full cycloplegic refraction). These glasses will be changed to reflect changes in refractive error or frame fit as appropriate at follow up.
  Arms: B1 (intervention); B2 (intervention)

SUMMARY:
This is a feasibility study to begin investigating the possibility that early use of near vision glasses will improve vision in infants at risk of Cerebral Visual Impairment (CVI), leading to further improvement in other areas of development. This active intervention, starting at either 2 or 4 months of age (depending on randomisation), could be more effective than waiting until a problem is detected before giving glasses.

As this is a feasibility study, the investigators are looking at a small sample of babies (n=75) to see whether their parents/carers are willing to take part in a 3-arm study comparing two differently timed interventions to a control group, as well as looking at different aspects of the research plan in preparation for a larger final study.

DETAILED DESCRIPTION:
The aim of this study is to assess the feasibility and the acceptability of randomisation and the intervention, namely near vision glasses, from parents of very young babies at risk of Cerebral Visual Impairment (CVI).

All infants are born with an immature visual system, and for vision to develop normally, a clear image needs to transmit to the visual centres of the brain.

Good vision plays an important role in facilitating normal development so if CVI goes unnoticed, it can have a damaging effect on the child's early development, and subsequent education and quality of life. Children use their sight to learn to walk, talk, think and communicate. For this reason, early intervention has the potential to have positive effects on children's vision and general development.

Previous studies have shown that up to 75% of school age children, who have CVI, have difficulty focussing their eyes on a near target, so near objects, such as their hands and parents' faces, will appear blurry. These studies also showed that wearing glasses for near focus improved vision but has not been assessed in babies.

This is a single-centre, parallel group, open-label feasibility trial to assess the feasibility of testing the effect near vision glasses (full cycloplegic refraction plus 3.00D add for near) could have on the visual and developmental outcome in babies at risk of brain injury.

Infants at risk of developing CVI include those who have had hypoxic ischaemic encephalopathy (HIE) and those born prematurely before 29 weeks gestation.

The paediatric research optometrist will enrol and assess all eligible babies of consenting families; first visit at 8 or 16 weeks corrected gestational age, depending on randomisation. Each infant will be followed up 3 months and 6-months (+/- 3 weeks) after the first visit.

There are three main areas of the assessment, which will be leading to potential primary outcome measures:

1. Visual Responses (including visual acuity and refractive status)

   At each visit, vision will be evaluated using Atkinson's battery for Child Development for Examining Functional Vision (ABCDEFV) according to the child's age and their ability. This comprises age-appropriate core vision tests (such as visual acuity and fixing and following) as well as additional tests that assess visual perception and visuomotor behaviour. If visual acuity cannot be obtained using Keeler acuity cards, as per ABCDEFV, the children will receive a measure using a Near Detection Scale (NDS).
2. General Development and Neurodevelopmental Delay

   Non-visual developmental assessments will include the Bayley Scales of Infant Development - 3rd edition (BSID-III) assessment as appropriate for age at routine neonatal clinical appointments at 3, 6,12 and 24 months (not the research clinics). A Prechtl video will also be performed at the 3-month appointment to assess the presence of fidgety movements. The presence of these movements at 3 months corrected gestational age has been strongly correlated with normal motor development.
3. Functional broadband near infrared spectroscopy (fBNIRS)

   i. Identification of changed functional haemodynamic and metabolic response to visual stimulus in infants at risk of visual dysfunction.

   ii. Assessment of changes in functional response in relation to response to glasses

   Eligible children with consenting parents will be screened for high refractive error prior to randomisation by the research optometrist to avoid post-randomisation dropouts. Evidence of high refractive error (more than -6.00D spherical equivalent or +8.00D spherical equivalent) will result in a referral to ophthalmology and exclusion from the study due to the possibility of associated ocular pathology with high refractive error.

   All of the above assessments have been organised at University College London Hospitals (UCLH). If the infant is randomised to get glasses, they will be given a near vision spectacle prescription (full cycloplegic refraction plus 3.00D add for near) to take to Great Ormond Street Hospital Eye Department dispensing optician to get the special glasses ordered.

   Expert ethical advice has been sought through the NIHR's Research Design Service to check on the dimension of potential harm (with a positive review). Each case will be monitored by the independent data monitoring and ethics committee (IDMEC) using follow up data who will report to the trial steering committee (TSC). The IDMEC, Trial Steering Committee (TSC) and Trial Management Group (TMG) will oversee the conduct of this trial.

ELIGIBILITY:
Inclusion criteria:

1. All term infants undergoing therapeutic hypothermia for hypoxic ischaemic encephalopathy (HIE).
2. All preterm infants born at <29 weeks gestational age.

Specifically, all children fulfilling these criteria will be eligible. Evidence of hypo-accommodation is not required.

Exclusion criteria:

1. Infants that are still an inpatient at 8 weeks corrected gestational age.
2. Ocular exclusion criteria: children with unrelated congenital or developmental ocular abnormality such as cataract requiring surgery, genetic retinal disease, coloboma. Retinopathy of prematurity will not be an exclusion criterion.
3. Infants with high refractive error (more than -6.00D spherical equivalent or +8.00D spherical equivalent).

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-06-09 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The acceptance of randomisation | 10 months
  This will be measured as the proportion of patients/parents who accept the offer of randomisation.

SECONDARY OUTCOMES:
Success rate in dispensing glasses to children in groups B1 and B2. | 6 months
  The percentage of infants dispensed vs. the total number of infants randomised to the intervention arms will be recorded at the end of the study.
Success rate of compliance with glasses for infants in groups B1 and B2. | 6 months
  The proportion of infants (%) who are still wearing their glasses at the 3 and 6 month follow-up appointments.
Visual Acuity | 6 months
  The distribution of visual acuity at the 3 and 6-month follow ups compared with visual acuity at the first visit in all 3 arms.
Retention rate | 15 months
  This will be measured by the median number of infants reported per month.
Refractive outcomes | 6 months
  The distribution of refractive outcomes (measured in dioptres) at 3 and 6-month follow ups as compared to the first visit in all 3 groups.
Evidence of impaired emmetropisation following administration of FMT | 6 months
  This will be measured by combining refractive error and visual acuity measures. The trial will not be feasible if there is a 2SD difference without compensatory benefit eg 2 lines improvement in visual acuity.
Determination of appropriate resource-use data collection methods | 15 months
  A targeted paediatric client service receipt inventory (CSRI) form has been designed specifically for this population and will be used for the duration of the feasibility study.
Accommodative outcomes | 6 months
  The distribution of accommodative outcomes (measured in dioptres) at 3 and 6-month follow ups as compared to the first visit in all 3 groups.
Completion of compliance questionnaires | 6 months
  Proportion of families completing phone questionnaire on spectacle compliance as a percentage of those in the intervention groups (B1 & B2).
Significant mechanical trauma | 6 months
  Significant mechanical trauma will be measured as the percentage of infants who have had an adverse event (from mechanical trauma) vs. the total number of infants prescribed glasses in groups B1 and B2. The study will not be feasible if this is more than 30% of infants in the intervention arms.
Consent rate | 10 months
  This will be measured as the number of infants recruited vs. number of infants, who fulfil the inclusion/exclusion criteria, approached.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom

REFERENCES:
- [Derived] Bullaj R, Dyet L, Mitra S, Bunce C, Clarke CS, Saunders K, Dale N, Horwood A, Williams C, St Clair Tracy H, Marlow N, Bowman R. Effectiveness of early spectacle intervention on visual outcomes in babies at risk of cerebral visual impairment: a parallel group, open-label, randomised clinical feasibility trial protocol. BMJ Open. 2022 Sep 21;12(9):e059946. doi: 10.1136/bmjopen-2021-059946. PMID 36130761